CLINICAL TRIAL: NCT04356469
Title: Study of TCR Alpha Beta T-Cell and CD19 B-Cell Depletion for Hematopoietic Cell Transplantation From Haploidentical Donors in the Treatment of Non-Malignant Hematological Disorders in Children
Brief Title: TCR Alpha Beta T-cell Depleted Haploidentical HCT in the Treatment of Non-Malignant Hematological Disorders in Children
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAP-HEM; IRB00249753 (Other: JHU ACH IRB)
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Hemoglobinopathy (Disorder); Severe Aplastic Anemia; Bone Marrow Failure Syndrome
MeSH Terms: conditions — Hemoglobinopathies; Anemia, Aplastic; Bone Marrow Failure Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TCR alpha beta T cell depletion (Experimental): The leukapheresis product will undergo TCR alpha beta negative selection following a standardized protocol
  Interventions: Biological: Haploidentical Hematopoietic Cell Transplantation

INTERVENTIONS:
Biological: Haploidentical Hematopoietic Cell Transplantation — TCR alpha beta T-cell and CD19 B-cell depleted haploidentical transplantation

SUMMARY:
This research is being done to learn if a new type of haploidentical transplantation using TCR alpha beta and CD19 depleted stem cell graft from the donor is safe and effective to treat the patient's underlying condition. This study will use stem cells obtained via peripheral blood or bone marrow from parent or other half-matched family member donor. These will be processed through a special device called CliniMACS, which is considered investigational.

ELIGIBILITY:
Inclusion Criteria:

1. Severe sickle cell disease (HbSS, HbSC, HbSB0, HbSB+, HbSD, HbSE) with at least one of the following criteria:

   1. Cerebrovascular accident lasting longer than 24 hours
   2. Impaired neuropsychological function with abnormal brain MRI/MRA
   3. Patients with frequent (≥ 3 per year for preceding 2 years) painful vaso-occlusive episodes
   4. Recurrent (≥ 3 in lifetime) acute chest syndrome events which have necessitated erythrocyte transfusion therapy
   5. Any combination of ≥ 3 acute chest syndrome episodes and vaso-occlusive pain episodes yearly for 3 years and have failed treatment with hydroxyurea (HU) (at least 6 months on maximum tolerated dose) or who are intolerant to HU therapy
2. Thalassemia major with at least one of the following criteria:

   1. Transfusion dependency defined as receiving 8 or more transfusions per year
   2. Thalassemia diagnosis documented by clinical assessment, laboratory evidence with microcytic anemia and absence of HbA (< 10%) on electrophoresis and or confirmation by DNA analysis of alpha and beta gene loci
   3. Genotypically proven thalassemia major for children < 2 years of age even in the absence of transfusion dependency
   4. Lucarelli class 1 or 2 risk status (i.e. with only 0-2 of the following factors: hepatomegaly, portal fibrosis, or poor response to chelation therapy)
3. Bone marrow failure syndromes and autoimmune cytopenias:

   1. Severe Aplastic Anemia refractory to immunosuppressive therapy
   2. Diamond Blackfan Anemia refractory to conventional therapy
   3. Inherited Bone Marrow Failure Syndromes such as Fanconi anemia and Shwachman-Diamond syndrome with progressive marrow failure (without cytogenetic evidence of MDS/AML)
   4. Severe Congenital Neutropenia
   5. Congenital Amegakaryocytic Thrombocytopenia
   6. Glanzmann Thrombasthenia
   7. Autoimmune Cytopenias refractory to conventional treatment (including Pure red cell aplasia, Evan's syndrome, Immune thrombocytopenia, autoimmune hemolytic anemia)
   8. Other marrow failure disorders not otherwise specified

Inclusion Criteria:

1. Patient has a suitable genotypic identical match of 5/10. The donor and recipient must be identical, as determined by high resolution typing, at least one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-C, HLA-DRB1 and HLA-DQB1.
2. Patients must have adequate organ function measured by:

   1. Cardiac: asymptomatic or if symptomatic then LVEF at rest must be ≥ 40% or SF ≥ 26%
   2. Pulmonary: asymptomatic or if symptomatic DLCO ≥ 40% of predicted (corrected for hemoglobin) or pulse oximetry ≥ 92% on room air if the patient is unable to perform pulmonary function testing.
   3. Renal: Creatinine clearance (CrCl) or glomerular filtration rate (GFR) must be > 50 mL/min/1.73 m2.
   4. Hepatic: Serum conjugated (direct) bilirubin < 2.0 x ULN for age as per local laboratory unless attributable to Gilbert's syndrome; AST and ALT < 5.0 x ULN for age as per local laboratory. Patients with hyperbilirubinemia as a consequence of hyperhemolysis, or a profound change in serum hemoglobin post blood transfusion, are not excluded.
   5. Karnofsky or Lansky (age-dependent) performance score ≥ 50
3. Signed written informed consent

Exclusion Criteria:

1. Participants who have an HLA-matched sibling who is able and willing to donate bone marrow. Patients with a HLA-matched unrelated donors are not excluded.
2. Pregnant or breastfeeding females.
3. Patient has HIV or uncontrolled fungal, bacterial or viral infections.
4. Patient has received prior solid organ transplant.
5. Patient has active GVHD (> grade II) or chronic extensive GVHD due to a previous allograft at the time of inclusion.
6. For patients with hemoglobinopathy, liver biopsy is necessary if the patient has received chronic transfusions for over a year and has two ferritin levels of ≥ 1000 ng/ml. Patients with cirrhosis, extensive bridging hepatic fibrosis, or active hepatitis are excluded from enrollment.

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Estimated)
Dates: Start 2020-07-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of successful donor engraftment | Day 100 after transplantation
  The incidence of engraftment at day 100 will be described based on donor chimerism in the whole blood and or fractions sorted for T-cell and myeloid subsets. The donor chimerism will be scored as autologous reconstitution (< 5% donor), mixed chimerism (5-49%=low mixed, 50-95%=high mixed), > 95%=full donor chimerism.

SECONDARY OUTCOMES:
Overall survival and Event-free survival | Up to 2 years post transplant
  Overall survival is defined as the time of enrollment to death from any cause or last follow up.
  Event-free survival is defined as the time of enrollment to death, primary or secondary graft failure, graft failure necessitating a second HCT procedure, DLI or stem cell boost given for treatment of falling chimerism, or disease recurrence
Kinetics of neutrophil and platelet engraftment | Up to 42 days post transplant
  Neutrophil engraftment defined as absolute neutrophil count ≥500/μL for 3 consecutive measurements on different days and platelet engraftment defined as sustained platelet count >20,000/μL and >50,000//μL with no platelet transfusions in the preceding seven days.
Transplant-related mortality | Up to 100 days post transplant
  Rate of transplant-related mortality
Acute grade II-IV GvHD and Chronic GvHD | Up to 2 years post transplant
  Incidence and severity of acute and chronic graft versus host disease
Primary and secondary graft failure | Up to 2 years post transplant
  Rates of primary and secondary graft failure
Transplant-related complications and infections | Up to 2 years post transplant
  Frequency of transplant-related complications and rate of infections following transplantation
Cellular and Immunological reconstitution by laboratory evaluations | Up to 2 years post transplant
  The recovery of different lymphocyte subpopulation (CD3+; CD4+; CD8+; CD3+CD45RA+and CD45RO; TCR alpha beta; TCR gamma delta; CD19+)

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Chellapandian, MD, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Johns Hopkins All Children's Hospital, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: No